CLINICAL TRIAL: NCT05172167
Title: Prospective Evaluation of Antibodies Levels Variation Against SARS-CoV-2 in a Vaccinated Population of the Metropolitan Area of Valle de Aburra . Pilot Prospective Cohort.
Brief Title: Prospective Evaluation of SARS-CoV-2 Antibodies Levels in a Vaccinated Population of Valle de Aburra
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Antioquia (Other)
Collaborators: Laboratorio integrado de medicina especializada(LIME) (Unknown); Proyecto de regalias BPIN 2020000100152 (Unknown)
Responsible Party: Principal Investigator, Andres Felipe Zuluaga Salazar, Full profesor, senior researcher and head of the Department of Pharmacology and Toxicology in Antioquia University, Universidad de Antioquia
Other Study IDs: LIME-21-P-02
Record Dates: First submitted 2021-12-23; First posted 2021-12-29 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: Laboratory biomarkers; Health condition; COVID-19; Antibodies level; Vaccinated people
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early vaccinated against COVID-19: 80 subjects with less than 4 months after being fully vaccinated against COVID-19
  Interventions: Diagnostic Test: Levels of IgG and IgM SARS-CoV-2 antibodies blood test.; Diagnostic Test: RT-PCR SARS-CoV-2 nasopharyngeal swab
- Late vaccinated against COVID-19: 80 subjects with more than 4 months after being fully vaccinated against COVID-19
  Interventions: Diagnostic Test: Levels of IgG and IgM SARS-CoV-2 antibodies blood test.; Diagnostic Test: RT-PCR SARS-CoV-2 nasopharyngeal swab
- COVID-19 infection: 40 patients diagnostic of COVID-19
  Interventions: Diagnostic Test: Levels of IgG and IgM SARS-CoV-2 antibodies blood test.; Diagnostic Test: RT-PCR SARS-CoV-2 nasopharyngeal swab

INTERVENTIONS:
Diagnostic Test: Levels of IgG and IgM SARS-CoV-2 antibodies blood test. — 0,1,2 months
Diagnostic Test: RT-PCR SARS-CoV-2 nasopharyngeal swab — 0,1,2 months

SUMMARY:
Recent research evidence shows that levels of antibodies acquierd post vacunation against SARS-Cov-2 decrease over time as well as the efficacy to control the infection, additionally in a multicenter study carried out in 2020 were evidenced differences in the time it took to decrease the antibodies according to the type of vaccine, defined as mRNA or other types of vaccine.

In this study , the variation of the SARS-Cov-2 antibody levels in patients from Valle de Aburrá will be correlated according to the COVID-19 vaccine received.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will undergo a serial IgM -IgG COVID-19 antibodies blood test and SARS-Cov-2 PCR by nasopharingeal swab, that will be taken at the beginning of the study and mensually for two months.

During the study will be done an active search for SARS-CoV-2 infections in the vaccinated people cohort, and if it is posible to characterize the variant of SARS-CoV-2 in participants previously vaccinated against this pathogen.

The main objective of this study is to describe the pattern of antibodies blood test based in the type of vaccine and correlated the pattern of antibodies SARS-Cov-2 levels in a population of Valle de Aburrá.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years old
* The vaccinated patients to be included must have received a complete vaccination scheme for COVID-19 according to the Ministerio de Salud y Protección Social de Colombia
* SARS-CoV-2 infection in the last 2 months, verified by rtPCR test

Exclusion Criteria:

* Immunocompromised patients
* Immunosuppressive treatments, chemotherapy or antiretroviral therapy
* Outpatient anticoagulant therapy
* For vaccinated people (groups 1 and 2): if have had COVID-19 infection in the last 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with a fully vaccination scheme for COVID-19 according to the Ministerio de Salud y Protección Social de Colombia and patients diagnosed with SARS-CoV-2 infection in the last 60 days, without matter vaccination status against SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
IgG and IgM antibodies blood test levels generated by the different COVID-19 vaccines in people throughout the time of the study. | Through study completion, an average of 2 months

SECONDARY OUTCOMES:
Comparing immunoglobulins M and G levels in vaccinated patients against SARS-CoV-2 with RNA and non RNA vaccines. | Through study completion, an average of 2 months
SARS-CoV-2 infections in vaccinated patients against COVID-19. | Through study completion, an average of 2 months
Correlate through time immunoglobulins M and G levels in people vaccinated against COVID-19 and SARS-CoV-2 acute infected patients. | Through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Andres F Zuluaga, MD, MSc, MeH, Principal Investigator — Universidad de Antioquia
Locations (1):
- Laboratorio Integrado de Medicina Especializada, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided